CLINICAL TRIAL: NCT03939130
Title: Effects of Fructose Rich Diet Associated With Aerobic Training on Uric Acid Levels and Endothelial Function
Brief Title: Fructose Rich Diet and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alvaro Reischak-Oliveira, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 84642318.8.0000.5347
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Fructose Metabolism Disorder; Fructose Rich Diet; Metabolic Disease; Aerobic Exercise
MeSH Terms: conditions — Metabolic Diseases | interventions — Fructose; Glucose; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fructose-rich diet (Experimental): Subjects will be submitted to a standard diet associated with a sweetened beverage (provided by the researchers) during 4 weeks. Without knowing the content (blind), they will receive fructose based beverage, prepared as a solution with 10% fructose, water and flavoring powder, totaling 1.0g / kg of body mass / day of fructose.
  Interventions: Dietary Supplement: Fructose
- Glucose-rich diet (Active Comparator): Subjects will be submitted to a standard diet associated with a sweetened beverage (provided by the researchers) during 4 weeks. Without knowing the content (blind), they will receive glucose based beverage, prepared as a solution with 10% glucose, water and flavoring powder, totaling 1.0g / kg of body mass / day of glucose.
  Interventions: Dietary Supplement: Glucose
- Fructose-rich diet and exercise (Experimental): The subjects will perform the same protocol described in the intervention Fructose-rich diet, except for the inclusion of the physical exercise. During the 4-week intervention, participants will perform three sessions a week of 60 minutes of aerobic exercise at 60% of VO2 peak on cycle ergometer.
  Interventions: Other: Fructose and exercise

INTERVENTIONS:
Dietary Supplement: Fructose — Consumption of 1.0g / kg of body mass / day of fructose.
  Arms: Fructose-rich diet
Dietary Supplement: Glucose — Consumption of 1.0g / kg of body mass / day of glucose.
  Arms: Glucose-rich diet
Other: Fructose and exercise — Consumption of 1.0g / kg of body mass / day of fructose + 3 weekly sessions of 60 minutes of aerobic exercise.
  Arms: Fructose-rich diet and exercise

SUMMARY:
Cardiometabolic diseases have been associated with high consumption of sweetened beverages. These products are responsible for the largest portion of the total consumption of fructose in the diet and it is suggested that excessive intake of this monosaccharide may contribute to the development of risk factors for these diseases due to differences in metabolism relative to glucose. However, there is a lack of data in the literature demonstrating the deleterious effects of excessive fructose consumption on vasodilation and whether aerobic training may be able to prevent or mitigate these damages in humans. Therefore, the aim of the study will be to verify the effect of 4 weeks of high fructose diet associated with aerobic training on uric acid levels and its influence on markers related to oxidative stress and vasodilatation. Twenty-one sedentary men and women, aged between 19 and 35 years, will be submitted to 4 weeks of intervention. In a randomized way, subjects will be divided into 3 groups: high fructose diet, high glucose diet and high fructose diet and exercise. Blood samples will be taken before, in the middle and after the intervention to verify the concentrations of uric acid, superoxide dismutase enzyme, thiobarbituric acid, nitrite / nitrate, lipid profile, glucose, insulin, C-reactive protein and endothelin-1. In addition, flow-mediated dilatation, insulin resistance index, pancreatic beta cell functional capacity index, oral glucose tolerance test, 24-hour blood pressure, heart rate variability and body composition will be analyzed. The comparisons will be performed through the Generalized Estimates of Equations, adopting the factors group and time. The Bonferroni post-hoc will be used to identify differences. The accepted level of significance will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* Not engaged in regular exercises;
* Aged between 19 and 35 years;
* Body mass index (BMI) of less than 30kg / m².

Exclusion Criteria:

* Individuals with BMI below 18kg / m² and greater than 30kg / m²;
* Smokers;
* Dyslipidemic;
* Diabetic;
* Hypertensive;
* Alcohol use;
* Appetite suppressants use;
* Medications use;
* Supplements use;
* Chronic disease that impedes the performance of physical exercise.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Flow Mediated Dilatation | 4 weeks
Concentration of Uric Acid | 4 weeks
Concentration of Nitrite / Nitrate | 4 weeks

SECONDARY OUTCOMES:
Concentration of Superoxide Dismutase Enzyme | 4 weeks
Concentration of Substances Reactive to Thiobarbituric Acid | 4 weeks
  Oxidative stress outcome
Concentration of Total Cholesterol | 4 weeks
Concentration of Triglycerides | 4 weeks
Concentration of Low-Density Lipoprotein | 4 weeks
Concentration of High-Density Lipoprotein | 4 weeks
Concentration of Glucose | 4 weeks
Concentration of Insulin | 4 weeks
HOMA-IR | 4 weeks
HOMA-B | 4 weeks
Insulin Sensitivity | 4 weeks
  Oral glucose tolerance test
Concentration of C-Reactive Protein | 4 weeks
Concentration of Endothelin-1 | 4 weeks
24-hour Blood Pressure | 4 weeks
Heart Rate Variability | 4 weeks
Body Fat | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No